CLINICAL TRIAL: NCT02149433
Title: Early Steroid Use in Infants With Clinical Pneumocystis Jiroveci Pneumonia (PCP) in the Queen Elizabeth Central Hospital, Blantyre, Malawi
Brief Title: Pneumocystis Jerovici Pneumonia in Infants and Steroids
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kamuzu University of Health Sciences (Other)
Responsible Party: Principal Investigator, Elizabeth Molyneux, Lecturer Paediatrics and Professor, Kamuzu University of Health Sciences
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: Pneumocystis and Steroids
Record Dates: First submitted 2012-07-09; First posted 2014-05-29 (Estimated); Last update posted 2015-12-11 (Estimated); Status verified 2015-12

CONDITIONS: Pneumonia, Pneumocystis Jerovici
Keywords: Pneumocystis Jiroveci; Steroids; Infants
MeSH Terms: conditions — Pneumonia | interventions — Prednisone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Prednisone versus placebo (Experimental): Prednisone 2mg/kg orally once a day x 7 days, 1 mg/kg orally once a day x 7 days and then 0.5 mg/kg orally once a day x 7 days
  Interventions: Drug: Prednisone; Drug: Placebo

INTERVENTIONS:
Drug: Prednisone — The steroid regime will be oral prednisone at 2 mg/kg for 7 days, then 1 mg/kg for 7 days, then 0.5mg/kg for 7 days for a total of 21 days.
Drug: Placebo

SUMMARY:
This is a double-blind randomized controlled trial assessing the efficacy of adjuvant corticosteroids in clinically diagnosed Pneumocystis jiroveci pneumonia in infants.

DETAILED DESCRIPTION:
The study aims to determine whether the early administration of adjuvant corticosteroids in addition to high dose oral Co-trimoxazole reduces mortality amongst infants aged 2-6 months with vertically acquired HIV and clinically diagnosed Pneumocystis jiroveci pneumonia. Infants will be randomized to receive either a steroid regime of oral prednisolone at 2 mg/kg for 7 days, then 1 mg/kg for 7 days, then 0.5mg/kg for 7 days for a total of 21 days or placebo.

ELIGIBILITY:
Inclusion Criteria:

* Consecutive infants with HIV and clinical features of Pneumocystis jiroveci pneumonia who require oxygen (oxygen saturations in air < 90%).
* Clinical diagnosis of Pneumocystis jiroveci pneumonia will be made by one of the study investigators. All infants must be HIV ELISA positive or exposed, have an oxygen requirement (saturations on air < 90%) and have severe respiratory distress and cough. They may also have a low grade fever, clear chest or diffuse signs on auscultation and features suggestive of Pneumocystis jiroveci infection on chest radiography.

Exclusion Criteria:

* Previous known allergy or hypersensitivity or other contraindication to corticosteroids or co-trimoxazole.
* Previous treatment for suspected Pneumocystis jiroveci pneumonia or a delay starting steroids for greater than 24 hours after starting high dose co-trimoxazole.
* Patients who are not exposed to HIV.
* Infants with known preexisting active pulmonary or cardiac disease.
* Patients who do not live within the Blantyre district and who are unable to attend follow up at QECH.
* Infants whose parents or guardians refuse consent.

Ages: 2 Months to 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 78 (Actual)
Dates: Start 2012-05; Primary Completion 2014-08 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Reduction in inpatient mortality by 20%. | 36 months
  To determine whether the addition of oral Prednisolone to standard treatment reduces inpatient mortality by 20% in patients aged 2-6 months with clinical PJP pneumonia.

SECONDARY OUTCOMES:
Commencement of antiretroviral treatment | 36 months
  To determine whether steroids significantly increase the number of patients that successfully commence anti-retroviral treatment.
6 month survival | 36 months
  To determine whether steroids significantly increase the number of patients that survive to 6 months following commencement of anti-retrovirals.
Morbidity (days in hospital and days on oxygen) | 36 months
  To determine whether steroids significantly alter morbidity as determined by number of days spent in hospital as an inpatient and number of days on oxygen.

CONTACTS AND LOCATIONS:
Overall Officials: Laura Newberry, MD, Principal Investigator — Paediatric Department, College of Medicine, University of Malawi; Elizabeth Molyneux, FRCPCH, Study Director — Paediatric Department, College of Medicine, University of Malawi
Locations (1):
- Queen Elizabeth Central Hospital, Blantyre, Malawi